CLINICAL TRIAL: NCT04641156
Title: Effect of Adding Supervised Physical Therapy Exercise Program to Photobiomodulation Therapy in the Treatment of Cervicogenic Somatosensory Tinnitus: A Randomized Controlled Study
Brief Title: Effect of Physical Therapy Exercise Program and Low-Level Laser Therapy on the Treatment of Cervicogenic Somatosensory Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, Professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6688
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low level LASER Therapy (Experimental): Subjects in this group received low-level laser therapy
  Interventions: Other: Exercise Therapy program added to laser therapy
- Exercise group (Experimental): Subjects in this group received additional planned exercise therapy program
  Interventions: Other: Exercise Therapy program added to laser therapy

INTERVENTIONS:
Other: Exercise Therapy program added to laser therapy — a supervised physical therapy exercise program for the neck muscles in the form of manual mobilizations for sternocleidomastoid muscle and upper fibers of trapezius in addition to myofascial trigger point release

SUMMARY:
To determine the effectiveness of adding a physical therapy exercise program to low-level laser therapy on the treatment of chronic tinnitus treatment

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 45 to 55 years old both sex
* Unilateral tinnitus
* Stable tinnitus for at least 3 months
* suffering from severe chronic non-fluctuating subjective cervicogenic somatic tinnitus (CST)

Exclusion Criteria:

* tinnitus with clear ontological etiologies as perforation of the tympanic membrane
* external otitis media
* conductive hearing loss
* patients with a traumatic cervical spine injury, tumors
* Any history of exposure to ototoxic drugs/substances
* psychotic disorders with auditory hallucination

Ages: 45 Years to 55 Years | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
VAS | 8 weeks
  Numerical estimates of tinnitus severity before and after treatment for both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt